CLINICAL TRIAL: NCT02839291
Title: Evaluation of Medical Practice in the Management of Bone Metastases After Injectable Bone Antiresorptive Treatment, and Its Influence on Quality of Life
Acronym: PRISM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2015/279
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Tumor With Bone Metastasis

ARMS (1):
- quality of life questionaries (Experimental): Patients should complete 3 quality of life questionaries (EORTC-QLQ C30 ; EORTC QLQ-BM22 and Euroqol EQ-5D) at many time points : at inclusion, every 3 months and at the end of study visit (2 years after inclusion)
  Interventions: Other: quality of life questionaries; Drug: intravenous or oral bone antiresorptive treatments

INTERVENTIONS:
Other: quality of life questionaries
Drug: intravenous or oral bone antiresorptive treatments

SUMMARY:
To evaluate the current medical practice and its influence on health-related quality of life, in patients who are treated with injectable bone antiresorptive drugs (biphosphonates or denosumab) for at least one year.

DETAILED DESCRIPTION:
This protocol will evaluate the pursuit of injectable bone antiresorptive treatments or their switch to oral biphosphonates, or treatment stop, in the contexte of medical practice.

The primary end-point is the health-related quality of life (QoL). Secondary endpoints are safety, overall survial, the impact of toxicities of the treatment on QoL, and the description of supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven tumor with bone metastasis, single or multiple (with or without metastasis extra-osseous)
* Patients treated with injectable bone antiresorptive therapy for 12 months or more
* Signed written informed consent

Exclusion Criteria:

* patient with any medical or psychiatric condition or disease which would make the patient inappropriate to complete quality of life questionaries
* patient under guardianship, curator or under the protection of justice, pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
evaluation of 4 targeted dimensions of the EORTC-QLQ-BM22 quality of life questionarie | to 6 months
  evaluation of 4 parameters: painful sites characteristics of pain, functional impairment, psychosocial aspect

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Hôpital Nord Franche-Comté, Montbéliard